CLINICAL TRIAL: NCT01994018
Title: Correlation Between Relapses in Multiple Sclerosis (MS) and Vitamin D Intake
Status: Completed | Type: Observational
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Reuben Valenzuela, Reuben Mari Valenzuela, MD, OSF Healthcare System
Other Study IDs: OSF-13-002
Record Dates: First submitted 2013-10-18; First posted 2013-11-25 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
Keywords: Vitamin D; Interferon Beta; Glatiramer Acetate; Relapse rates
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control Group (Vitamin D level): Twenty (20) healthy individuals not on vitamin D supplementation will be used as controls to get a baseline vitamin D level.
- MS Group: RR-MS patients treated with a FDA approved immuno-modulatory drug with and without vitamin D supplementation for at least 2 years.
- Retrospective Chart Review: RR-MS patients treated with a FDA approved immuno-modulatory drug for MS.

SUMMARY:
The correlation between relapses in MS and vitamin D intake will be examined.

DETAILED DESCRIPTION:
Research suggests that a connection between vitamin D and MS could be tied to the positive effects vitamin D has on the immune system. Published data also shows a synergistic effect of vitamin D in conjunction with Glatiramer acetate (GA), an already approved FDA immunomodulating drug, in the treatment of multiple sclerosis. Further correlation of vitamin D and GA or Interferon Beta needs to be tested.

This is a retrospective pilot study in which 100 patients diagnosed with relapsing-remitting MS (RR-MS) according to the McDonald criteria and treated with either GA or interferon with and without vitamin D supplementation for at least 2 years were included. Only RR-MS patients who received FDA approved immuno-modulatory drugs for MS are included in this review.

Relapses before and during treatment will be analyzed and a subgroup analysis will be done on those who received vitamin D and those who did not. Magnetic resonance Imaging (MRI) of the brain and cervical spine of these MS patients will also be reviewed to see if there is any correlation between radiologic changes, relapses and vitamin D level.

The 100 MS patients involved the chart review will be invited to participate in a one time blood draw to measure vitamin D levels. Additionally, the MS patients will be asked about their relapse status and medication history.

Twenty (20) healthy individuals not on vitamin D supplementation will be used as controls to get a baseline vitamin D level.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria (MS Group):

  * Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
  * Be age 18 or older at the time of informed consent.
  * Have a diagnosis of relapsing-remitting multiple sclerosis (RR-MS) as defined by the McDonald Criteria.
  * Are taking FDA approved immune-modulatory drugs for MS.
  * Patients had at least one relapse during the year prior to initiation of MS treatment.
  * After at least 2 years on therapy, patients were classified as MS responders (MS-R) or MS non-responders (MS-NR) based on a clinical criteria recently reported in the literature. A responder (MS-R) is a patient with an annual relapse rate (ARR) < 0.5 and no evidence of disease progression as measured by EDSS (expanded disability status scale). A hypo/non-responder (MS-NR) is a patient with an ARR > 0.5 and/or with progression in the EDSS of at least 1 point sustained for 6 months.

Inclusion Criteria (Control Group):

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Be age 18 or older at the time of informed consent.
* Have not taken any vitamin D supplementation for more than 12 months.

Exclusion Criteria:

* Exclusion Criteria (MS Group):

  * Those who have a diagnosis of secondary progressive MS (SPMS) or primary progressive MS (PPMS).
  * Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol.
  * Any other condition, clinical finding, or reason that, in the opinion of the Investigator, is determined to be unsuitable for enrollment into this study.
  * Those who received other forms of treatment under than a FDA approved MS drugs are excluded.

Exclusion Criteria(Control Group):

* Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol.
* History of osteoporosis, kidney disease, parathyroid disease, problems with calcium metabolism, sacrcoidosis, and/or pregnancy.
* Current nursing home or bed bound patients.
* Any other condition, clinical finding, or reason that, in the opinion of the Investigator, is determined to be unsuitable for enrollment into this study.

Inclusion Criteria (Retrospective Chart Review) • Only RR-MS patients who received FDA approved immuno-modulatory drugs for MS.

Exclusion Criteria (Retrospective Chart Review)

• Patients diagnosed with MS sub-types other than RR-MS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MS Group: Relapsing-remitting MS (RR-MS) patients according to the McDonald criteria who are treated with a FDA approved immuno-modulatory drugs.
  Control Group: Healthy individuals not on vitamin D supplementation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
• Annual relapse rates | After at least 2 years on therapy with an approved immuno-modulatory drug for MS.
  Data collected from retrospective chart review part of study

SECONDARY OUTCOMES:
Expanded Disability Status Scale | After at least 2 years on therapy with an approved immuno-modulatory drug for MS.
  Data collected from retrospective chart review part of study.
Multiple Sclerosis Responders | After at least 2 years on therapy with an approved immuno-modulatory drug for MS.
  Data collected from retrospective chart review part of study.
Multiple Sclerosis Non-Responders | After at least 2 years on therapy with an approved immuno-modulatory drug for MS.
  Data collected from retrospective chart review part of study.
Response to immunodulators among patients who received MS treatment with or without vitamin D | After at least 2 years on therapy with an approved immuno-modulatory drug for MS.
  Data collected from retrospective chart review part of study.
non-response to immunodulators among patients who received MS treatment with or without vitamin D | After at least 2 years on therapy with an approved immuno-modulatory drug for MS.
  Data collected from retrospective chart review part of study.
MRI (brain images) | after at least 2 years on therapy with an approved immuno-modulatory drug for MS.
  Data collected from retrospective chart review part of study.

OTHER OUTCOMES:
Serum Vitamin D levels in subjects taking GA with Vitamin D supplementation. | Within 30 days of consent or when patient is able
Serum Vitamin D levels in subjects taking GA without Vitamin D supplementation | Within 30 days of consent or when patient is able
Serum vitamin D levels in subjects taking Interferon Beta with vitamin D supplementation | Within 30 days of consent or when patient is able
Serum vitamin D levels in subjects taking Interferon Beta without vitamin D supplementation | Within 30 days of consent or when patient is able
serum vitamin D levels from the control group | Within 30 days of consent or when patient is able

CONTACTS AND LOCATIONS:
Overall Officials: Reuben M Valenzuela, MD, Principal Investigator — OSF Healthcare System
Locations (1):
- OSF Saint Francis Medical Center, Peoria, Illinois, United States

REFERENCES:
- [Background] D'hooghe MB, Haentjens P, Nagels G, Garmyn M, De Keyser J. Sunlight exposure and sun sensitivity associated with disability progression in multiple sclerosis. Mult Scler. 2012 Apr;18(4):451-9. doi: 10.1177/1352458511423778. Epub 2011 Sep 27. PMID 21952096
- [Background] Smolders J, Moen SM, Damoiseaux J, Huitinga I, Holmoy T. Vitamin D in the healthy and inflamed central nervous system: access and function. J Neurol Sci. 2011 Dec 15;311(1-2):37-43. doi: 10.1016/j.jns.2011.07.033. Epub 2011 Aug 23. PMID 21862439
- [Background] O'Connor K, Weinstock-Guttman B, Carl E, Kilanowski C, Zivadinov R, Ramanathan M. Patterns of dietary and herbal supplement use by multiple sclerosis patients. J Neurol. 2012 Apr;259(4):637-44. doi: 10.1007/s00415-011-6226-3. Epub 2011 Sep 6. PMID 21898138
- [Background] Weinstock-Guttman B, Zivadinov R, Ramanathan M. Inter-dependence of vitamin D levels with serum lipid profiles in multiple sclerosis. J Neurol Sci. 2011 Dec 15;311(1-2):86-91. doi: 10.1016/j.jns.2011.07.024. Epub 2011 Aug 16. PMID 21849177
- [Background] McDowell TY, Amr S, Culpepper WJ, Langenberg P, Royal W, Bever C, Bradham DD. Sun exposure, vitamin D intake and progression to disability among veterans with progressive multiple sclerosis. Neuroepidemiology. 2011;37(1):52-7. doi: 10.1159/000329258. Epub 2011 Aug 5. PMID 21822026